CLINICAL TRIAL: NCT05410730
Title: Phase I/II Clinical Study of Dose Escalation and Dose Expansion of SHR-1501 Alone or in Combination With Bacille de Calmette Guerin （BCG） or SHR-1316 in the Treatment of Non-muscle Invasive Bladder Cancer（NMIBC）
Brief Title: A Study of SHR-1501 Alone or in Combination With BCG or SHR-1316 in Subjects With NMIBC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1501-I-103
Record Dates: First submitted 2022-05-19; First posted 2022-06-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-07

CONDITIONS: High-risk NMIBC

STUDY DESIGN:
Intervention Model Description: Single Group .Dose escalation and expansion of SHR-1501 alone or in combination with BCG or SHR-1316 in the treatment of NMIBC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1501 (Experimental): * Phase I：Phase Ia and Ib： Phase Ia include SHR-1501 dose escalation and expansion; Phase Ib ： SHR-1501 in combination with BCG or SHR-1316 dose escalation
  * Phase II：SHR-1501 in combination with BCG or SHR-1316 dose expansion in NMIBC
  Interventions: Drug: SHR-1501

INTERVENTIONS:
Drug: SHR-1501 — SHR-1501 single agent dose escalation, and in combination of BCG or SHR-1316.

SUMMARY:
The study is to evaluate the safety and tolerability of SHR-1501 alone or in combination with BCG or SHR-1316 in the patients with NMIBC, and to determine the RP2D of SHR-1501 in combination with BCG or SHR-1316.

To evaluate the preliminary efficacy of SHR-1501 alone or in combination with BCG or SHR-1316 in the treatment of NMIBC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study, understand the research procedures and be able to sign the informed consent in writing;
2. Age ≥ 18 years old, gender is not limited;
3. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
4. Expected survival time ≥ 2 years;
5. High-risk NMIBC diagnosed by previous pathological biopsy
6. Cystoscopy within 6 weeks before the first administration shows that the lesion has been completely removed, or the residual lesion is only carcinoma in situ; for T1 stage lesions, postoperative pathological results must show the presence of bladder muscle tissue;
7. ineligible or unwilling to undergo radical cystectomy;
8. The level of organ function is good.
9. use contraceptive measures (such as intrauterine device and contraceptive pill) during the study treatment period and within 3 months after the end of the study treatment period, and the female subject and the female partner of the male subject should use highly effective contraceptive methods; the female subject of childbearing age without surgical sterilization must be negative for serum HCG within 7 days before the first administration and must be non-lactating.

Exclusion Criteria:

1. Received surgery or radiotherapy for bladder lesions within 2 weeks before the first administration;
2. Those who have previously received the following treatments and have not experienced disease progression before enrolment t as assessed by the investigator:

   * Intravesical instillation of cytotoxic chemotherapy or other drugs;
   * Immune checkpoint inhibitor;
   * Other investigational products for the treatment of NMIBC.
3. Currently receiving study treatment in other clinical trials or less than 4 weeks from last participation to the first administration of this study;
4. Upper urinary tract tumor detected by CTU or MRU during screening period, urethral prostate tumor detected by cystoscopy, or other concomitant malignant tumors within 5 years before the first administration;
5. Previous medical history or examination suggests active tuberculosis within 1 year prior to the first dose;
6. Serious infection within 4 weeks before the first administration, or undefined fever>38.5 ℃ during screening/before the first administration;
7. Obvious urinary tract infections and gross hematuria, indicating safety issues assessed by the investigators;
8. Patients who discontinued treatment due to adverse reactions such as toxemia, systemic infection or urinary incontinence during previous BCG treatment;
9. Using of immunosuppressive drugs within 2 weeks prior to the first administration, excluding nasal and inhaled corticosteroids, low physiological doses of systemic steroids, and prophylactic anti allergic steroids;
10. Active or history of interstitial lung disease;
11. History of clinically significant cardiovascular disease
12. A history of immunodeficiency, including HIV seropositive, other acquired or congenital immunodeficiency diseases, a history of organ transplantation, or those who are using immunosuppressants;
13. With a history of active autoimmune disease；
14. Patient with active hepatitis B (HBeAg positive and HBV DNA ≥ 500 IU/mL), hepatitis C (HCV antibody positive and HCV RNA higher than the detection limit of the analytical method);
15. Known allergic or intolerance to study drug, BCG (Phase Ib and Phase II subjects only) or excipients;
16. The presence of other serious physical or mental illness, abnormal laboratory tests, and other factors that may increase the risk of participating in the study, or interfere with the results of the study; and any other conditions that the investigator deems inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 21 Days
Maximum tolerated dose | Approximately 2years
Recommended Phase 2 dose (RP2D) | Approximately 2 years.
CR Rate (cohort 2) | Approximately 4 years.
12-month DFS Rate (cohort 1、3、4) | Approximately 4 years

SECONDARY OUTCOMES:
Treatment-Related Adverse Events as assessed by CTCAE v5.0 | Approximately 4 years.
Duration of CR (DoR) | Approximately 4 years.
CR rate at 6 months and 18 months | Approximately 4 years.
DFS | Approximately 4 years.
Time to cystectomy, | Approximately 4 years.
Radical cystectomy rate; | Approximately 4 years.
The amount of drug recovered in perfusate and urine after SHR-1501 perfusion | Approximately 5 years.
Maximum concentration (Cmax) of SHR-1501 | Approximately 2 years, if applicable
Time to maximum concentration (Tmax) of SHR-1501 | Approximately 2 years，if applicable
Areas under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of SHR-1501 | Approximately 2 years，if applicable
Areas under the concentration-time curve from time zero extrapolated to infinity (AUCinf) of SHR-1501 | Approximately 2 years，if applicable
Half-life (t1/2) of SHR-1501 | Approximately 2 years, if applicable
Apparent clearance (CL/F) of SHR-1501 | Approximately 2 years, if applicable
Apparent volume of distribution (V/F) of SHR-1501 | Approximately 2 years, if applicable
Concentration of SHR-1501 in Urine | Approximately 2 years, if applicable
Anti-drug antibody of SHR-1501 | Approximately 2 years
Neutralizing antibody of SHR-1501 | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided